CLINICAL TRIAL: NCT02265705
Title: A Randomized, Double-Blind, Placebo-Controlled, Phase 3 Study Evaluating the Efficacy and Safety of Baricitinib in Patients With Moderately to Severely Active Rheumatoid Arthritis Who Have Had an Inadequate Response to Methotrexate Therapy
Brief Title: A Study of Baricitinib (LY3009104) in Participants With Rheumatoid Arthritis (RA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14875; I4V-CR-JAGS (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-10-13; First posted 2014-10-16 (Estimated); Results first posted 2019-03-13 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — baricitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Baricitinib (Experimental): 4 milligrams (mg) baricitinib administered orally once a day for 52 weeks. Participants with renal impairment will receive 2 mg baricitinib orally once a day for 52 weeks.
  Participants will continue to take background methotrexate (MTX) therapy throughout study. Other background therapies, including non-steroidal anti-inflammatory drugs (NSAIDs) and low dose oral corticosteroids, are permitted during the study for participants who are on stable doses of these treatments at baseline.
  Interventions: Drug: Baricitinib
- Placebo (Placebo Comparator): Placebo administered orally once a day through week 24. At week 24, participants will be given 4 mg or 2 mg (participants with renal impairment) baricitinib orally once a day through Week 52.
  Participants will continue to take background MTX therapy throughout study. Other background therapies, including NSAIDs and low dose oral corticosteroids, are permitted during the study for participants who are on stable doses of these treatments at baseline.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Baricitinib — Administered orally
  Other Names: LY3009104; INCB 028050
  Arms: Baricitinib
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the safety and effectiveness of the study drug known as baricitinib in participants with moderately to severely active rheumatoid arthritis who have had an inadequate response to methotrexate therapy.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of adult-onset RA as defined by the ACR/European League Against Rheumatism (EULAR) 2010 Criteria for the Classification of RA.
* Have moderately to severely active RA defined as the presence of at least 6/68 tender joints and at least 6/66 swollen joints.
* Have a CRP (or hsCRP) measurement ≥ 6 mg/liter (L) based on the most recent data (if available).
* Have had regular use of MTX for at least the 12 weeks prior to study entry at a dose that, in accordance with local clinical practice, is considered acceptable to adequately assess clinical response. The dose of MTX must have been a stable, unchanging oral dose of 7.5 to 25 mg/week (or the equivalent injectable dose) for at least the 8 weeks prior to study entry. The dose of MTX is expected to remain stable throughout the study and may be adjusted only for safety reasons.

Exclusion Criteria:

* Are currently receiving corticosteroids at doses >10 mg of prednisone per day (or equivalent) or have been receiving an unstable dosing regimen of corticosteroids within 2 weeks of study entry or within 6 weeks of planned randomization.
* Have started treatment with NSAIDs within 2 weeks of study entry or within 6 weeks of planned randomization or have been receiving an unstable dosing regimen of NSAIDs within 2 weeks of study entry or within 6 weeks of planned randomization.
* Are currently receiving concomitant treatment with MTX, hydroxychloroquine, and sulfasalazine or combination of any 3 conventional disease modifying anti-rheumatic drugs (cDMARDs).
* Are currently receiving or have received cDMARDs (for example, gold salts, cyclosporine, azathioprine, or any other immunosuppressives) other than MTX, hydroxychloroquine (up to 400 mg/day), or sulfasalazine (up to 3000 mg/day) within 8 weeks prior to study entry.
* Have received leflunomide in the 12 weeks prior to study entry (or within 4 weeks prior to study entry if the standard 11 days of cholestyramine is used to washout leflunomide).
* Have started a new physiotherapy treatment for RA in the 2 weeks prior to study entry.
* Have ever received any biologic DMARD (such as tumor necrosis factor (TNF), interleukin-1, interleukin-6 (IL-6), or T-cell- or B-cell-targeted therapies).
* Have received any parenteral corticosteroid administered by intramuscular or intravenous injection within 2 weeks prior to study entry or within 6 weeks prior to planned randomization or are anticipated to require parenteral injection of corticosteroids during the study.
* Have had 3 or more joints injected with intraarticular corticosteroids or hyaluronic acid within 2 weeks prior to study entry or within 6 weeks prior to planned randomization.
* Have a diagnosis of any systemic inflammatory condition other than RA such as, but not limited to, juvenile chronic arthritis, spondyloarthropathy, Crohn's disease, ulcerative colitis, psoriatic arthritis, active vasculitis or gout.
* Have an estimated glomerular filtration rate (eGFR) based on the most recent available serum creatinine using the Modification of Diet in Renal Disease (MDRD) method of <40 milliliters/minute/1.73 meters squared (m^2).
* Have a history of chronic liver disease with the most recent available aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >1.5 times the upper limit of normal (ULN) or the most recent available total bilirubin 1.5 times the ULN.
* Have a current or recent (<30 days prior to study entry) clinically serious viral, bacterial, fungal, or parasitic infection.
* Have a history of active hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV).
* Have had household contact with a person with active tuberculosis (TB) and did not receive appropriate and documented prophylaxis for TB.
* Have evidence of active TB or have previously had evidence of active TB and did not receive appropriate and documented treatment.
* Are pregnant or nursing at the time of study entry.
* Are females of childbearing potential who do not agree to use 2 forms of highly effective birth control when engaging in intercourse while enrolled in the study and for at least 28 days following the last dose of orally administered investigational product.
* Are males who do not agree to use 2 forms of highly effective birth control while engaging in sexual intercourse with female partners of childbearing potential while enrolled in the study and for at least 28 days following the last dose of orally administered investigational product.
* Have previously been randomized in this study or any other study investigating baricitinib.
* Have received prior treatment with an oral janus kinase inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2014-10; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (22):
- Argentina (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ciudad Autonoma de Buenos Aire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rosario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Miguel de Tucumán
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., São Paulo, Brazil
- China (17):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beijing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bengbu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Changsha
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chengdu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guangzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hefei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jinan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kunming
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nanjing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ningbo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pingxiang
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shanghai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shantou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tianjin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wuhan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yancheng
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zhuzhou

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Taylor PC, Takeuchi T, Burmester GR, Durez P, Smolen JS, Deberdt W, Issa M, Terres JR, Bello N, Winthrop KL. Safety of baricitinib for the treatment of rheumatoid arthritis over a median of 4.6 and up to 9.3 years of treatment: final results from long-term extension study and integrated database. Ann Rheum Dis. 2022 Mar;81(3):335-343. doi: 10.1136/annrheumdis-2021-221276. Epub 2021 Oct 27. PMID 34706874
- [Derived] Yang Y, Xu J, Xu J, Li X, Hu J, Li X, Zhang X, He D, Bao C, Li Z, Wang G, Zerbini CAF, Spindler AJ, Kannowski CL, Wu H, Ji F, Zhan L, Liu M, Li Z. Patient-reported outcomes from a randomized, double-blind, placebo controlled, phase III study of baricitinib versus placebo in patients with moderately to severely active rheumatoid arthritis and an inadequate response to methotrexate therapy: results from the RA-BALANCE study. Ther Adv Musculoskelet Dis. 2021 Apr 20;13:1759720X211006964. doi: 10.1177/1759720X211006964. eCollection 2021. PMID 33959198
- [Derived] Li ZG, Hu JK, Li XP, Yang Y, Li XF, Xu JH, Zhang X, Xu J, Bao CD, He DY, Li ZJ, Wang GC, Zuo XX, Liu Y, Xiao ZY, Chen JW, Xin XF, Li JY, Jiang LD, Liu MR, Ji F, Li CG. Rapid Onset of Efficacy of Baricitinib in Chinese Patients with Moderate to Severe Rheumatoid Arthritis: Results from Study RA-BALANCE. Adv Ther. 2021 Jan;38(1):772-781. doi: 10.1007/s12325-020-01572-y. Epub 2020 Nov 25. PMID 33237533
- [Derived] Yang Y, Li XF, Zhang X, Bao CD, Hu JK, Xu JH, Li XP, Xu J, He DY, Li ZJ, Wang GC, Wu HJ, Ji F, Zhan LJ, Zerbini CAF, Li ZG. Efficacy and Safety of Baricitinib in Chinese Rheumatoid Arthritis Patients and the Subgroup Analyses: Results from Study RA-BALANCE. Rheumatol Ther. 2020 Dec;7(4):851-866. doi: 10.1007/s40744-020-00231-6. Epub 2020 Sep 2. PMID 32876903

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who did not respond (nonresponders) to study drug were eligible for rescue treatment (Tx) beginning at Week 16.
  Nonresponders were defined as lack of improvement of at least 20% in both tender joint count and swollen joint count at both Weeks 14 and 16 compared to baseline.
Groups:
- Placebo Treatment Period Week 0-24; Placebo Follow-up Period: Placebo administered orally once a day through week 24. At week 24, participants will be given 4 mg or 2 mg (participants with renal impairment) baricitinib orally once a day through Week 52.
- 4 Milligrams (mg) Baricitinib Treatment Period Week 0-24; 4 mg Baricitinib Treatment Period Week 24-52; 4 mg Baricitinib Follow-up Period: 4 mg baricitinib administered orally once a day for 52 weeks. Participants with renal impairment will receive 2 mg baricitinib orally once a day for 52 weeks.
- Rescue Treatment Period Week 16-52: All participants who are non-responders (both baricitinib and placebo arms) will receive rescue therapy at Week 16.
- Placebo to Baricitinib Treatment Period Week 24 - 52: At week 24, participants will be given 4 mg or 2 mg (participants with renal impairment) baricitinib orally once a day through Week 52.
Period: Treatment Period Week 0-24
Arm/Group | Placebo Treatment Period Week 0-24 | 4 Milligrams (mg) Baricitinib Treatment Period Week 0-24 | Rescue Treatment Period Week 16-52 | Placebo to Baricitinib Treatment Period Week 24 - 52 | 4 mg Baricitinib Treatment Period Week 24-52 | Placebo Follow-up Period | 4 mg Baricitinib Follow-up Period
Started | 145 | 145 | 0 | 0 | 0 | 0 | 0
Received at Least One Dose of Study Drug | 145 | 145 | 0 | 0 | 0 | 0 | 0
Rescued | 59 | 17 | 0 | 0 | 0 | 0 | 0
Completed | 133 ("Completers" include rescued participants.) | 136 ("Completers" include rescued participants.) | 0 | 0 | 0 | 0 | 0
Not Completed | 12 | 9 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Entry Criteria Not Met | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 5 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Rescue Period
Arm/Group | Placebo Treatment Period Week 0-24 | 4 Milligrams (mg) Baricitinib Treatment Period Week 0-24 | Rescue Treatment Period Week 16-52 | Placebo to Baricitinib Treatment Period Week 24 - 52 | 4 mg Baricitinib Treatment Period Week 24-52 | Placebo Follow-up Period | 4 mg Baricitinib Follow-up Period
Started | 0 (Participants who were nonresponders based on tender/swollen joint count entered into rescue group.) | 0 (Participants who were nonresponders based on tender/swollen joint count entered into rescue group.) | 77 (Participants who were determined to be nonresponders based on tender/swollen joint count.) | 0 | 0 | 0 | 0
Completed | 0 | 0 | 74 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 3 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Open Label Period
Arm/Group | Placebo Treatment Period Week 0-24 | 4 Milligrams (mg) Baricitinib Treatment Period Week 0-24 | Rescue Treatment Period Week 16-52 | Placebo to Baricitinib Treatment Period Week 24 - 52 | 4 mg Baricitinib Treatment Period Week 24-52 | Placebo Follow-up Period | 4 mg Baricitinib Follow-up Period
Started | 0 | 0 | 0 | 74 (Completed Wk 24 w/o rescue Tx, switched to or remained on active Tx, and entered Open Label Period.) | 120 (Completed Wk 24 w/o rescue Tx, switched to or remained on active Tx, and entered Open Label Period.) | 0 | 0
Completed | 0 | 0 | 0 | 72 | 115 | 0 | 0
Not Completed | 0 | 0 | 0 | 2 | 5 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 2 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 2 | 0 | 0
Period: Follow-up Period
Arm/Group | Placebo Treatment Period Week 0-24 | 4 Milligrams (mg) Baricitinib Treatment Period Week 0-24 | Rescue Treatment Period Week 16-52 | Placebo to Baricitinib Treatment Period Week 24 - 52 | 4 mg Baricitinib Treatment Period Week 24-52 | Placebo Follow-up Period | 4 mg Baricitinib Follow-up Period
Started | 0 | 0 | 0 | 0 | 0 | 2 (Participants from placebo who never rescued or switched and entered post-treatment follow-up period.) | 58 (Participants who ever took baricitinib and entered the post-treatment follow-up period.)
Completed | 0 | 0 | 0 | 0 | 0 | 1 | 47
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 11
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 0 | 1 | 6
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-Treat (mITT) population includes all randomized participants who received at least one dose of the study drug.
Groups:
- Placebo: Placebo administered orally once a day through week 24. At week 24, participants will be given 4 mg or 2 mg (participants with renal impairment) baricitinib orally once a day through Week 52.
  Participants will continue to take background MTX therapy throughout study. Other background therapies, including NSAIDs and low dose oral corticosteroids, are permitted during the study for participants who are on stable doses of these treatments at baseline.
  Placebo: Administered orally
- Baricitinib: 4 milligrams (mg) baricitinib administered orally once a day for 52 weeks. Participants with renal impairment will receive 2 mg baricitinib orally once a day for 52 weeks.
  Participants will continue to take background methotrexate (MTX) therapy throughout study. Other background therapies, including non-steroidal anti-inflammatory drugs (NSAIDs) and low dose oral corticosteroids, are permitted during the study for participants who are on stable doses of these treatments at baseline.
  Baricitinib: Administered orally
- Total: Total of all reporting groups
Arm/Group | Placebo | Baricitinib | Total
Number analyzed (Participants) | 145 | 145 | 290
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (12.7) | 49.5 (10.6) | 49.2 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106 | 127 | 233
  Male | 39 | 18 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 115 | 116 | 231
  Unknown or Not Reported | 30 | 29 | 59
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 5 | 6
  Asian | 115 | 116 | 231
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 26 | 24 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 22 | 21 | 43
  China | 115 | 116 | 231
  Brazil | 8 | 8 | 16
Duration of Rheumatoid Arthritis [Mean (Standard Deviation); unit: years] — Time from symptom onset of Rheumatoid Arthritis.
  years | 9.1 (7.0) | 10.7 (8.3) | 9.9 (7.7)
Tender Joint Count of 68 Evaluable Joints [Mean (Standard Deviation); unit: Tender Joints] — TJC is the number of tender and painful joints determined for each participant by examination of 68 joints. Joints were assessed by pressure and joint manipulation on physical examination. Participants were asked for pain sensations on these manipulations and watched for spontaneous pain reactions. Any positive response on pressure, movement, or both was translated into a single tender-versus-nontender dichotomy.
  Tender Joints | 25.2 (14.7) | 23.3 (13.6) | 24.2 (14.2)
Swollen Joint Count of 66 Evaluable Joints [Mean (Standard Deviation); unit: Swollen Joints] — SJC is the number of swollen joints determined for each participant by examination of 66 joints. Joints were classified as either swollen or not swollen. Swelling was defined as palpable fluctuating synovitis of the joint.
  Swollen Joints | 14.8 (9.5) | 14.6 (8.6) | 14.7 (9.1)
High Sensitivity C-Reactive Protein (hsCRP) [Mean (Standard Deviation); unit: milligrams per liter (mg/L)] — hsCRP is a laboratory analyte that is an indicator of inflammation. Decreases in hsCRP represent reductions in inflammation.
  milligrams per liter (mg/L) | 26.48 (31.27) | 25.59 (23.53) | 26.04 (27.63)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving 20% Improvement in American College of Rheumatology Criteria (ACR20)
Description: ACR20 Responder Index is a composite of clinical, laboratory, and functional measures in rheumatoid arthritis (RA). An ACR20 Responder is a participant who had ≥20% improvement from baseline in both 68 tender and 66 swollen joint counts and ≥20% improvement in at least 3 of 5 criteria: Patient's and Physician's Global Assessment of Disease Activity, Health Assessment Questionnaire-Disability Index (HAQ-DI) (assessment of participant's physical function), pain due to RA, and hsCRP. Participants who discontinue before analysis time point are treated as non-responders. Percentage of participants achieving ACR20 response = (number of ACR20 responders) / (number of participants analyzed) * 100.
Time Frame: Week 12
Population: All randomized participants who received at least one dose of the study drug.
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Placebo administered orally once a day through week 24. At week 24, participants will be given 4 mg or 2 mg (participants with renal impairment) baricitinib orally once a day through Week 52.
- Baricitinib: 4 mg baricitinib administered orally once a day for 52 weeks. Participants with renal impairment will receive 2 mg baricitinib orally once a day for 52 weeks.
Arm/Group | Placebo | Baricitinib
Number analyzed (Participants) | 145 | 145
percentage of participants | 28.3 | 58.6
Statistical Analysis 1: Comparison: Placebo vs Baricitinib; Test type: Superiority; p = 0.001, Regression, Logistic; Odds Ratio (OR) = 4.1, 95% CI 2-sided [2.5 to 6.9]

2. Secondary Outcome: Change From Baseline to Week 12 in the Health Assessment Questionnaire Disability Index (HAQ-DI) Score
Description: The HAQ-DI questionnaire assesses the participant's self-perception on the degree of difficulty [0 (without any difficulty), 1 (with some difficulty), 2 (with much difficulty), and 3 (unable to do)] when dressing and grooming, arising, eating, walking, hygiene, reaching, gripping, and performing other daily activities. Scores for each functional area were averaged to calculate HAQ-DI scores, which ranged from 0 (no disability) to 3 (worst disability). A decrease in HAQ-DI score indicated an improvement in the participant's condition.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose of the study drug and had an evaluable score at Week 12.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Baricitinib
Number analyzed (Participants) | 145 | 144
units on a scale | -0.35 (0.52) | -0.57 (0.54)
Statistical Analysis 1: Comparison: Placebo vs Baricitinib; Test type: Superiority; p = 0.001, ANCOVA; Mean Difference (Final Values) = -0.20, 95% CI 2-sided [-0.31 to -0.09], Standard Error of Mean 0.056

3. Secondary Outcome: Change From Baseline to Week 12 in Disease Activity Score Modified to Include the 28 Diarthroidal Joint Count (DAS28)-High Sensitivity C-Reactive Protein (hsCRP)
Description: Disease Activity Score (DAS) modified to include 28 joint count (DAS28) consisted of composite score of following variables: tender joint count-28 (TJC28), swollen joint count-28 (SJC28), CRP (mg/L), and Patient's Global Assessment of Disease Activity using VAS (patient's global VAS). DAS28-CRP=0.56*square root (sqrt)(TJC28)+0.28*sqrt(SJC28)+0.36*natural log(CRP+1)+0.014*patient's global VAS+0.96. Scores ranged from 1.0-9.4, where lower scores indicated less disease activity, and remission was DAS28-CRP <2.6. A decrease in DAS28-CRP indicated an improvement in participant's condition.
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose of study drug and had an evaluable score at Week 12.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Baricitinib
Number analyzed (Participants) | 144 | 144
units on a scale | -0.94 (1.04) | -1.89 (1.14)
Statistical Analysis 1: Comparison: Placebo vs Baricitinib; Test type: Superiority; p = 0.001, ANCOVA; Mean Difference (Final Values) = -1.02, 95% CI 2-sided [-1.25 to -0.79], Standard Error of Mean 0.116

4. Secondary Outcome: Proportion of Participants Achieving a Simplified Disease Activity Index (SDAI) Score < or Equal to 3.3
Description: SDAI is a tool for measurement of disease activity in RA that integrates TJC28, SJC28, acute phase response using C-reactive protein (milligrams per liter), Participant's Global Assessment of Disease Activity using VAS centimeters (cm), and Physician's Global Assessment of Disease Activity using VAS (cm). The SDAI is calculated by summing the values of the 5 components. Lower scores indicated less disease activity. An index-based definition of remission occurs with an SDAI score ≤3.3.
Time Frame: Week 12
Population: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Baricitinib
Number analyzed (Participants) | 145 | 145
Participants | 0 | 2
Statistical Analysis 1: Comparison: Placebo vs Baricitinib; Test type: Superiority; Difference in response rate = 1.4, 95% CI 2-sided [-0.5 to 3.3]

5. Secondary Outcome: Median Duration of Morning Joint Stiffness in the 7 Days Prior to Week 12
Description: Participants recorded the duration of their morning joint stiffness (MJS) in hours and minutes into paper diaries daily. If morning joint stiffness duration was longer than 12 hours (720 minutes), it was truncated to 720 minutes for statistical presentations and analyses. The average value across the 7 days preceding each visit was calculated. A decrease in duration of morning joint stiffness indicated an improvement in the participant's condition.
Time Frame: Week 12
Population: All randomized participants who received at least one dose of study drug and had an evaluable score at Week 12.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Placebo | Baricitinib
Number analyzed (Participants) | 145 | 144
minutes | 47.6 [30.0 to 67.9] | 24.3 [15.0 to 30.6]
Statistical Analysis 1: Comparison: Placebo vs Baricitinib; Test type: Superiority; p = 0.004, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -12.9, 95% CI 2-sided [-28.0 to -2.9]

6. Secondary Outcome: Mean Severity of Morning Joint Stiffness in the 7 Days Prior to Week 12
Description: Participants rated the severity of their morning joint stiffness by selecting a number from 0 to 10 that best described their overall level of morning joint stiffness from the time they woke up, where 0 represents "no joint stiffness" and 10 represents "joint stiffness as bad as you can imagine". Participants reported their severity daily in paper diaries. The average value across the 7 days preceding each visit was calculated.
Time Frame: Week 12
Population: All randomized participants who received at least one dose of study drug and had an evaluable score at Week 12.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Baricitinib
Number analyzed (Participants) | 145 | 144
units on a scale | 4.3 (2.3) | 3.5 (2.1)
Statistical Analysis 1: Comparison: Placebo vs Baricitinib; Test type: Superiority; p = 0.002, ANCOVA; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.2 to -0.3], Standard Error of Mean 0.23

7. Secondary Outcome: Mean Worst Tiredness Numeric Rating Scale (NRS) in the 7 Days Prior to Week 12
Description: Participants rated their tiredness by selecting a number from 0 to 10 that best described their worst tiredness during the last 24 hours, where 0 represents "no tiredness" and 10 represents "as bad as you can imagine". Participants reported their worst tiredness in paper diaries. The average value across the 7 days preceding each visit is calculated.
Time Frame: Week 12
Population: All randomized participants who received at least one dose of study drug and had an evaluable score at Week 12.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Baricitinib
Number analyzed (Participants) | 145 | 144
units on a scale | 4.4 (2.0) | 3.7 (1.9)
Statistical Analysis 1: Comparison: Placebo vs Baricitinib; Test type: Superiority; p = 0.001, ANCOVA; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.2 to -0.4], Standard Error of Mean 0.20

8. Secondary Outcome: Mean Worst Pain NRS in the 7 Days Prior to Week 12
Description: Participants rated their joint pain by selecting a number from 0 to 10 that best described their worst joint pain during the last 24 hours, where 0 represents "no pain" and 10 represents "pain as bad as you can imagine". Participants reported their worst joint pain in daily paper diaries. The average value across the 7 days preceding each visit was calculated.
Time Frame: Week 12
Population: All randomized participants who received at least one dose of study drug and had evaluable score at Week 12.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Baricitinib
Number analyzed (Participants) | 145 | 144
units on a scale | 5.0 (1.8) | 4.1 (1.9)
Statistical Analysis 1: Comparison: Placebo vs Baricitinib; Test type: Superiority; p = 0.001, ANCOVA; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-1.3 to -0.5], Standard Error of Mean 0.20

ADVERSE EVENTS:
Time Frame: Start of treatment to end of study (Up To 52 Weeks)
Description: All randomized participants who received at least one dose of the study drug.
Arm/Group | Placebo Treatment Period Week 0-24 | 4 Milligrams (mg) Baricitinib Treatment Period Week 0-24 | Rescue Treatment Period Week 16-52 | Placebo to Baricitinib Treatment Period Week 24 - 52 | 4 mg Baricitinib Treatment Period Week 24-52 | Placebo Follow-up Period | 4 mg Baricitinib Follow-up Period
All-Cause Mortality (participants affected / at risk) | 0/145 | 0/145 | 1/77 | 0/74 | 0/120 | 0/2 | 0/58
Serious Adverse Events (participants affected / at risk) | 4/145 | 4/145 | 3/77 | 7/74 | 3/120 | 0/2 | 1/58
Other Adverse Events (participants affected / at risk) | 72/145 | 94/145 | 38/77 | 31/74 | 41/120 | 0/2 | 3/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo Treatment Period Week 0-24 (N=145) | 4 Milligrams (mg) Baricitinib Treatment Period Week 0-24 (N=145) | Rescue Treatment Period Week 16-52 (N=77) | Placebo to Baricitinib Treatment Period Week 24 - 52 (N=74) | 4 mg Baricitinib Treatment Period Week 24-52 (N=120) | Placebo Follow-up Period (N=2) | 4 mg Baricitinib Follow-up Period (N=58)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertrophic anal papilla (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/106 (0) | 1/127 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal tubular acidosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo Treatment Period Week 0-24 (N=145) | 4 Milligrams (mg) Baricitinib Treatment Period Week 0-24 (N=145) | Rescue Treatment Period Week 16-52 (N=77) | Placebo to Baricitinib Treatment Period Week 24 - 52 (N=74) | 4 mg Baricitinib Treatment Period Week 24-52 (N=120) | Placebo Follow-up Period (N=2) | 4 mg Baricitinib Follow-up Period (N=58)
Anaemia (Blood and lymphatic system disorders) | 14 (18) | 12 (13) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2) | 3 (4) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (10) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (2) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 5 (5) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Asthenia (General disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 6 (9) | 10 (11) | 6 (6) | 4 (6) | 4 (5) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 22 (24) | 28 (37) | 7 (8) | 5 (5) | 11 (12) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 5 (5) | 13 (14) | 10 (11) | 4 (4) | 3 (3) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 9 (11) | 5 (5) | 5 (5) | 2 (2) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 4 (4) | 5 (5) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 8 (9) | 16 (16) | 6 (6) | 3 (3) | 9 (9) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 4 (5) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (9) | 0 (0) | 2 (5) | 1 (1) | 3 (3) | 0 (0) | 3 (3)
Joint swelling (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 5 (7) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 8 (20) | 5 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0/22 (0) | 1/14 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 9 (9) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 8 (8) | 7 (7) | 4 (4) | 3 (4) | 6 (6) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-12-07): https://cdn.clinicaltrials.gov/large-docs/05/NCT02265705/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-12): https://cdn.clinicaltrials.gov/large-docs/05/NCT02265705/SAP_001.pdf